CLINICAL TRIAL: NCT05535244
Title: A Phase I/II, Open-Label, Multi-Cohort Study to Evaluate the Efficacy and Safety of Cevostamab in Prior B Cell Maturation Antigen-Exposed Patients With Relapsed/Refractory Multiple Myeloma
Brief Title: A Study Evaluating the Efficacy and Safety of Cevostamab in Prior B Cell Maturation Antigen (BCMA)-Exposed Participants With Relapsed/Refractory Multiple Myeloma
Acronym: CAMMA 2
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CO43476; 2021-006816-10 (EudraCT Number)
Record Dates: First submitted 2022-08-24; First posted 2022-09-10 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort A1: Prior BCMA antibody-drug conjugate (ADC) or chimeric antigen receptor T (CAR-T) (Experimental): Participants in Cohort A1 will be treated at the double step-up split dosing regimen.
  Interventions: Drug: Cevostamab; Drug: Tocilizumab
- Cohort A2: Prior BCMA Bispecific (Experimental): Participants enrolled into exploratory Cohort A2 will receive the same dosing regimen as Cohort A1.
  Interventions: Drug: Cevostamab; Drug: Tocilizumab
- Cohort B1: Prior BCMA CAR-T (Experimental): Participants enrolled in expansion Cohort B1, will be given cevostamab at the selected dosing regimen.
  Interventions: Drug: Cevostamab; Drug: Tocilizumab
- Cohort B2: Prior BCMA Bispecific (Experimental): Expansion Cohort B2 will be opened, after the initial results from Cohort A2, at the same dose as per Cohort B1.
  Interventions: Drug: Cevostamab; Drug: Tocilizumab

INTERVENTIONS:
Drug: Cevostamab — Cevostamab will be administered by IV infusion in 21-day cycles.
Drug: Tocilizumab — Tocilizumab will be administered for the treatment of cytokine release syndrome (CRS) when necessary.

SUMMARY:
This study will evaluate the efficacy, safety, and pharmacokinetics of cevostamab in participants with relapsed or refractory multiple myeloma (R/R MM) via intravenous (IV) infusion.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of MM based on standard International Myeloma Working Group (IMWG) criteria
* Evidence of progressive disease based on investigators determination of response by IMWG criteria on or after their last dosing regimen
* Prior BCMA ADC or CAR-T Cohort: participants who have received a BCMA-targeted CAR-T or ADC therapy and are triple-class relapsed or refractory
* Prior BCMA Bispecific Cohort: participants who have received a BCMA-targeting T-cell-dependent bispecific (TDB) antibody and are triple-class relapsed or refractory
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Life expectancy is at least 12 weeks
* Agreement to protocol-specified assessments, including bone marrow biopsy and aspirate samples as detailed in the protocol
* Resolution of AEs from prior anti-cancer therapy to Grade =< 1
* For female participants of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraception during the treatment period and for at least 5 months after the final dose of cevostamab and for 3 months after the last dose of tocilizumab was administered
* For male participants: agreement to remain abstinent (refrain from heterosexual intercourse) or use a condom, and agree to refrain from donating sperm during the treatment period and for at least 2 months after the final dose of tocilizumab (if applicable) to avoid exposing the embryo

Exclusion Criteria:

* Inability to comply with protocol-mandated hospitalization
* Pregnancy or breastfeeding, or intention of becoming pregnant during the study or within 5 months after the final dose of cevostamab or tocilizumab or within 3 months after the last dose of tocilizumab (if applicable)
* Prior treatment with cevostamab or another agent with the same target
* Prior BCMA ADC or CAR-T Cohort: prior treatment with any T cell dependent bi-specific antibody (TDB) antibody including non BCMA targeting TDB
* Prior use of any monoclonal antibody (mAb), radioimmunoconjugate, or ADC as anti-cancer therapy within 4 weeks before first study treatment, except for the use of non-myeloma therapy
* Prior treatment with systemic immunotherapeutic agents
* Prior treatment with CAR-T cell therapy within 12 weeks before first cevostamab infusion
* Known treatment-related, immune-mediated adverse events associated with prior checkpoint inhibitors
* Treatment with radiotherapy, any chemotherapeutic agent, or treatment with any other anti-cancer agent within 4 weeks or 5 half-lives of the drug, whichever is shorter, prior to first study treatment
* Autologous stem cell transplantation (SCT) within 100 days prior to first study treatment
* Prior allogeneic SCT
* Circulating plasma cell count exceeding 500/ microliter (µL) or 5% of the peripheral blood white cells
* Prior solid organ transplantation
* History of autoimmune disease
* History of confirmed progressive multifocal leukoencephalopathy
* History of severe allergic or anaphylactic reactions to mAb therapy
* Known history of amyloidosis
* Lesions in proximity of vital organs that may develop sudden decompensation/deterioration in the setting of a tumor flare
* History of other malignancy within 2 years prior to screening, except those with negligible risk of metastasis or death, such as ductal carcinoma in situ not requiring chemotherapy, appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, low-grade, localized prostate cancer not requiring treatment or appropriately treated Stage I uterine cancer
* Current or past history of central nervous system (CNS) disease, such as stroke, epilepsy, CNS vasculitis, neurodegenerative disease, or CNS involvement by MM
* Significant cardiovascular disease that may limit a potential participant's ability to adequately respond to a cytokine release syndrome (CRS) event
* Symptomatic active pulmonary disease or requiring supplemental oxygen
* Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection at study enrollment, or any major episode of infection requiring treatment with IV (intravenous) antimicrobials where the last dose of IV antimicrobial was given within 14 days prior to first study treatment
* Active symptomatic COVID-19 infection at study enrollment or requiring treatment with IV antiviral where the last dose of IV antiviral treatment was given within 14 days prior to first study treatment. Participants with active COVID-19 infection must have clinical recovery and two negative antigen tests at least 24 hours apart prior to first study treatment
* Positive and quantifiable Epstein-Barr virus (EBV) polymerase chain reaction (PCR) or cytomegalovirus (CMV) PCR prior to first study treatment
* Known or suspected chronic active EBV infection
* Known history of Grade >=3 CRS or immune effector cell-associated neurotoxicity syndrome (ICANS) with prior bispecific therapies
* Known history of hemophagocytic lymphohistiocytosis (HLH) or macrophage activation syndrome (MAS)
* Recent major surgery within 4 weeks prior to first study treatment
* Positive serologic or PCR test results for acute or chronic hepatitis B virus (HBV) infection
* Acute or chronic hepatitis C virus (HCV) infection
* Known history of human immunodeficiency virus (HIV) seropositivity
* Administration of a live, attenuated vaccine within 4 weeks before first study treatment or anticipation that such a live attenuated vaccine will be required during the study
* Treatment with systemic immunosuppressive medications, with the exception of corticosteroid treatment <= 10 mg/day prednisone or equivalent, within 2 weeks prior to first study treatment
* History of illicit drug or alcohol abuse within 12 months prior to screening, in the investigator's judgment
* Any medical condition or abnormality in clinical laboratory tests that, in the investigator's judgment, precludes the participant's safe participation in and completion of the study, or which could affect compliance with the protocol or interpretation of results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-10-17 (Actual); Primary Completion 2027-02-26 (Estimated); Study Completion 2027-02-26 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) as Determined by the Investigator | Baseline up to approximately 2 years
Percentage of Participants with Adverse Events | Baseline up to approximately 2 years

SECONDARY OUTCOMES:
ORR as Determined by the Independent Review Committee (IRC) | Baseline up to approximately 2 years
Duration of Response (DOR) | Baseline up to approximately 2 years
Rate of Complete Response (CR) or Better | Baseline up to approximately 2 years
Rate of Very Good Partial Response (VGPR) or Better | Baseline up to approximately 2 years
Overall Survival (OS) | Baseline up until death from any cause (up to approximately 2 years)
Progression-free Survival (PFS) | Baseline up to approximately 2 years
Time to First Response (for Participants who Achieve an Objective Response) | Baseline up to approximately 2 years
Time to Best Response (for Participants who Achieve an Objective Response) | Baseline up to approximately 2 years
Percentage of Participants Experiencing a Clinically Meaningful Improvement in the Fatigue Domain of the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Core-30 Questionnaire (QLQ-C30) and EORTC QLQ-MY20 | Baseline up to approximately 2 years
Time to Deterioration in the Fatigue Domain of the EORTC QLQ-C30 and/or Disease Symptoms Domain of the EORTC QLQ-MY20 | Baseline up to approximately 2 years
Serum Concentration of Cevostamab at Specified Timepoints | At Cycles 1, 2, 3, 4, 6, 8 and every other cycle until the end of treatment up to approximately 2 years. Each cycle is 21-days.
Number of Anti-drug Antibody (ADAs) Against Cevostamab at Baseline | Baseline
Percentage of Participants with ADAs Against Cevostamab During the Study | Up to approximately 2 years
Cytokine Release Syndrome (CRS) Following Administration of Tocilizumab | Baseline up to approximately 2 years
Relationship Between Serum Concentration of Cevostamab and Cytokine Release | Baseline up to approximately 2 years
Relationship Between Serum Concentration of Cevostamab and T Cell Number | Baseline up to approximately 2 years
Relationship Between Serum Concentration of Cevostamab and T-cell Activation State | Baseline up to approximately 2 years

OTHER OUTCOMES:
Minimal Residual Disease (MRD) Negative Rate | Baseline up to approximately 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (26):
- United States (8):
  - University of Colorado, Aurora, Colorado
  - Mayo Clinic-Jacksonville, Jacksonville, Florida
  - University of Maryland Greenebaum Cancer Center, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Tennessee Oncology - Nashville, Nashville, Tennessee
  - Hunstman Cancer Institute, Salt Lake City, Utah
- Australia (2):
  - Calvary Mater Newcastle, Waratah, New South Wales
  - St Vincent's Hospital Melbourne, Fitzroy, Victoria
- UZ Leuven Gasthuisberg, Leuven, Belgium
- France (3):
  - CHU NANTES - Hôtel Dieu, Nantes
  - APHP - Hospital Saint Louis, Paris
  - CHU de Poitiers - La Miletrie, Poitiers
- Germany (3):
  - Klinik der Uni zu Köln, Cologne
  - Universitätsklinikum Hamburg-Eppendorf Onkologisches Zentrum Medizinische Klinik II, Hamburg
  - Universitätsklinikum Würzburg, Würzburg
- Israel (3):
  - Hadassah Ein Karem Hospital, Jerusalem
  - Sheba Medical Center, Ramat Gan
  - Sourasky Medical Centre, Tel Aviv
- Italy (4):
  - Policlinico S.Orsola-Malpighi, Bologna, Emilia-Romagna
  - Asst Papa Giovanni Xxiii, Bergamo, Lombardy
  - Fond. IRCCS Istituto Nazionale Tumori, Milan, Lombardy
  - A.O. Città della Salute e della Scienza D - Osp. S. Giov. Battista Molinette, Turin, Piedmont
- Spain (2):
  - Hospital Clínic i Provincial, Barcelona
  - Hospital Univ. 12 de Octubre, Madrid

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing